CLINICAL TRIAL: NCT05525130
Title: Experimental Study of the Administration of a Food Supplement Containing Hydroxycitric Acid Versus Placebo in Patients With Oxalate and Calcium Phosphate Lithiasis in Whom Extracorporeal Shock Wave Lithotripsy is Indicated.
Brief Title: Study of the Administration of a Food Supplement in Patients With Lithiasis Treated With Extracorporeal Shock Wave Lithotripsy.
Acronym: FAGOTRICIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arafarma Group, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ARA-EXP/FAG-2019-03
Record Dates: First submitted 2022-06-07; First posted 2022-09-01 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Lithiasis; Nephrolithiasis
MeSH Terms: conditions — Lithiasis; Nephrolithiasis | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Food supplement (Experimental): Two doses (sachets) a day during 4 weeks before the ESWL. After the ESWL, one dose a day during 6 weeks.
  Interventions: Dietary Supplement: Food supplement
- Placebo (Placebo Comparator): Two doses (sachets) a day during 4 weeks before the ESWL. After the ESWL, one dose a day during 6 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Food supplement — FagolitosPlus® is an authorized food supplement that contains hydroxycitric acid, vitamin complexes and ions.
  Arms: Food supplement
Dietary Supplement: Placebo — Placebo has a composition that makes the weight and organoleptic characteristics are identical to FagolitosPlus®.
  Arms: Placebo

SUMMARY:
The extracorporeal shock wave lithotripsy (ESWL) is the treatment of choice for most stones in any of their locations. It is about breaking the stone without surgically intervening on the patient and getting him to expel the fragments himself.

It is thought that additional treatments to the ESWL could improve the success rate of ESWL for less favorable stones.

The components of our authorized food supplement have shown an inhibitory effect in vitro on the growth of calcium oxalate monohydrate crystals, even in hightly supersaturared solutions. Also these components show an inhibitory effect on the growth of calcium phosphate crystals. To sum up, it reduces the formation, inhibits the growth and promotes the dissolution of calcium oxalate and calcium phosphate kidney stones.

This is the reason why this experimental study aims to modify the size limit of the stones in the ESWL with adjuvant food supplement.

DETAILED DESCRIPTION:
The study treatment will be administered for 10 weeks. First, one dose will be administered every 12 hours for each patient during the 4 weeks prior to ESWL. After ESWL, and for 6 weeks, one dose will be administered every 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Renal lithiasis with high radiological and clinical suspicion of calcium oxalate or calcium phosphate, size of the largest diameter between 1.5x1cm and 2x1cm, which will be treated by ESWL, being symptomatic with little probability of spontaneous expulsion.
* Signed informed consent to participate in the clinical study.

Exclusion Criteria:

* Lithiasis of more than 20 mm and less than 15 mm for the largest diameter.
* Taking medications with influence on urinary lithogenesis (citrate, bicarbonate, thiazides, bisphosphonates, magnesium, calcium, vitamin B6, vitamin D, vitamin A, xanthine-oxidase inhibitors, uricosurics, probiotics, urease inhibitors, cystine binders, topiramate , antiretrovirals).
* Taking medications that influence urine pH (citrate, bicarbonate, carbonic anhydrase inhibitors, L-methionine, vitamin C, ammonium chloride).
* Taking selective serotonin reuptake inhibitor antidepressant medications.
* Taking anticoagulants and antiaggregants.
* ESWL contraindications: urine infection, active or recurrent; hemorrhagic diathesis; pregnant or lactating patients; others (extreme obesity, arterial aneurysm near the location of the stone, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2020-04-22 (Actual); Primary Completion 2022-09-16 (Actual); Study Completion 2022-10-05 (Actual)

PRIMARY OUTCOMES:
Efficacy of extracorporeal shock wave lithotripsy (ESWL) measured as reduction of the size (area) of lithiasis between both treatment groups. | 10 weeks after baseline visit
  To assess the level of fragmentation of lithiasis which is treated with ESWL by measuring the % of reduction of the size (area) of lithiasis through imaging tests.
Efficacy of extracorporeal shock wave lithotripsy (ESWL) measured as number of generated fragments between both treatment groups. | 10 weeks after baseline visit
  To assess the level of fragmentation of lithiasis which is treated with ESWL by measuring the number of generated fragments through imaging tests.
Efficacy of extracorporeal shock wave lithotripsy (ESWL) measured as the hardness of lithiasis between both treatment groups. | 10 weeks after baseline visit
  To assess the level of fragmentation of lithiasis which is treated with ESWL by measuring the hardness of lithiasis through imaging tests.

SECONDARY OUTCOMES:
Rate of morbidities related to the ESWL between both treatment groups. | 2 weeks and 6 weeks after ESWL
  All episodes of morbidities related to the ESWL will be recorded, whether considered relevant.

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Arrabal Martín, Dr, Study Chair — Hospital Universitario Clínico San Cecilio
Locations (3):
- Spain (3):
  - Hospital Universitario Clínico San Cecilio, Granada
  - Hospital Universitario Regional de Málaga, Málaga
  - Hospital Universitario Virgen de Valme, Seville

IPD SHARING:
Plan to Share IPD: Undecided